CLINICAL TRIAL: NCT03295955
Title: Comparing Efficacy of Postoperative Antibiotic Use in Transoral Thyroidectomy: a Prospective Randomized Controlled Trial Study
Brief Title: Comparing Efficacy of Postoperative Oral Antibiotic Use in Trans-Oral Thyroidectomy
Acronym: POTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Wook Yi, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1708-028-875
Record Dates: First submitted 2017-09-20; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Surgical Wound Infection; Thyroid Nodule
MeSH Terms: conditions — Surgical Wound Infection; Thyroid Nodule | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postop antibiotics group (Active Comparator): Prescribe Amoxicillin Clavulanate
  Interventions: Drug: Amoxicillin Clavulanate
- No postop antibiotics (No Intervention): Do not prescribe Amoxicillin Clavulanate

INTERVENTIONS:
Drug: Amoxicillin Clavulanate — Per-oral "Amoxicillin Clavulanate" Given or Non-given, after surgery
  Arms: Postop antibiotics group

SUMMARY:
Transoral endoscopic thyroid surgery is a emerging surgical technique for thyroid surgery. This study to investigate the need for postoperative antibiotics in transoral endoscopic thyroid surgery.

DETAILED DESCRIPTION:
To prevent possible infection from the oral cavity flora, most surgeons prescribe postoperative oral antibiotics more than 3 to 7 days after surgery. Currently, there's no clinical evidence that postoperative oral antibiotics is necessary or not in transoral endoscopic thyroid surgery. The investigator will conduct randomization after transoral thyroid surgery with two groups : postoperative oral antibiotics group versus no oral antibiotics group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who planned to Transoral endoscopic thyroidectomy
* Age between 20 to 70
* Voluntarily consenting to the study and study agreement
* No local invasion or distant metastasis
* Normal vocal cord function in laryngoscopic exam
* No significant abnormalities in preoperative laboratory tests

Exclusion Criteria:

* Take aspirin or antiplatelet drugs within 7 days before admission
* Uncontrolled hypertension, diabetes, chronic renal failure, or coagulation disease
* History of cardiovascular disease (angina pectoris, heart failure, myocardial infarction, history of coronary artery disease, stroke, transient ischemic attack)
* Substance abuse and alcohol abuse
* History of esophageal and airway diseases
* Patient was participated in other clinical trials within 30 days
* History of neck irradiation or surgery
* History of drug allergies
* Pregnant or lactating women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-03 (Estimated); Study Completion 2018-12-03 (Estimated)

PRIMARY OUTCOMES:
"CDC 1992 SSI table" score | Postoperative 1 day
  Clinical evidence of Surgical Site Infection
CBC, CRP | Postoperative 1 day
  Laboratory test

SECONDARY OUTCOMES:
Change of "CDC 1992 SSI table" score | Compare the CDC 1992 SSI table score between postoperative 1 day and 2 day/2 weeks.
  Clinical evidence of Surgical Site Infection
Change of CBC, CRP | Compare the CBC, CRP between postoperative 1 day and 2 day
  Laboratory test

CONTACTS AND LOCATIONS:
Locations (1):
- Jin Wook Yi, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Anuwong A, Ketwong K, Jitpratoom P, Sasanakietkul T, Duh QY. Safety and Outcomes of the Transoral Endoscopic Thyroidectomy Vestibular Approach. JAMA Surg. 2018 Jan 1;153(1):21-27. doi: 10.1001/jamasurg.2017.3366. PMID 28877292
- [Result] Anuwong A. Transoral Endoscopic Thyroidectomy Vestibular Approach: A Series of the First 60 Human Cases. World J Surg. 2016 Mar;40(3):491-7. doi: 10.1007/s00268-015-3320-1. PMID 26546193
- [Derived] Yi JW, Kim SJ, Lee KE. Evaluation of the efficacy of postoperative antibiotic treatment in transoral endoscopic thyroidectomy: a prospective randomised controlled trial. Br J Oral Maxillofac Surg. 2020 Apr;58(3):334-340. doi: 10.1016/j.bjoms.2020.01.004. Epub 2020 Jan 22. PMID 31982170